CLINICAL TRIAL: NCT04968262
Title: Urinary Actin, as a Potential Marker of Sepsis-related Acute Kidney Injury: a Pilot Study
Brief Title: Urinary Actin, as a Potential Marker of Sepsis-related Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dániel Ragán, MD, Principal Investigator, University of Pecs
Other Study IDs: no. 4327.316-2900/KK15/2011; KA-2018-17 (Other Grant/Funding Number: Medical School, University of Pécs)
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Sepsis; Acute Kidney Injury Due to Sepsis
Keywords: Sepsis-3; Acute Kidney Injury; Urinary actin; Western blot
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood; Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Patients receive sepsis therapy.
  Interventions: Other: Sepsis therapy
- Sepsis-related acute kidney injury: Patients receive sepsis and sepsis-related acute kidney injury therapy.
  Interventions: Other: Sepsis-related acute kidney injury therapy

INTERVENTIONS:
Other: Sepsis therapy — Patients receiving sepsis therapy followed the international guidelines of the 2016 Surviving Sepsis Campaign regarding fluid resuscitation, feeding, vasopressor, respiratory, anticoagulation and hydrocortisone therapy, along with ulcer prophylaxis and sedation. Blood and urine samples were collected at the intensive care unit from this patient group at three time points (T1-3): T1: within 24 hours after admission; T2: second day morning; T3: third day morning of follow-up. 24 patients were documented without sepsis and acute kidney injury as a control group.
  Groups: Sepsis
Other: Sepsis-related acute kidney injury therapy — Patient management of sepsis and sepsis-related acute kidney injury followed the international guidelines of the 2016 Surviving Sepsis Campaign regarding fluid resuscitation, feeding, vasopressor, respiratory, anticoagulation and hydrocortisone therapy, along with ulcer prophylaxis, sedation and renal replacement therapy (if needed). In this patient group, blood and urine sampling was performed at three time points (T1-3): T1: within 24 hours after admission; T2: second day morning; T3: third day morning of follow-up.
  Groups: Sepsis-related acute kidney injury

SUMMARY:
In our study, 17 septic, 43 sepsis-related acute kidney injury and 24 control patients were enrolled. Blood and urine samples were collected at the intensive care unit from acutely diagnosed septic and sepsis-related acute kidney injury patients at three time points (T1-3): T1: within 24 hours after admission; T2: second day morning; T3: third day morning of follow-up. Patients with malignancies needing palliative care, end-stage renal disease or kidney transplantation were excluded. Not more than one sample (venous blood, midstream spot urine) was collected from control patients. Serum and urinary actin levels were determined by quantitative Western blot. Urinary actin concentrations were expressed as µg/L, while serum actin levels were expressed as mg/L. Data were compared with laboratory and clinical parameters. Patients were categorized by the Sepsis-3 definitions and 30-day mortality data were investigated.

DETAILED DESCRIPTION:
Actin is a globular protein present in every cell with a 42 kilodalton molecular mass. It plays an important role in muscle contraction while being an essential component of the cytoskeleton as well. Several proteins (e.g. gelsolin, Gc-globulin) bind actin in the circulation during the physiological cell turnover, thus making its urinary appearance unlikely. However, recent studies indicate that actin could be detected in the urine of kidney-transplant patients with acute kidney injury. Therefore, the main focus of our research was the detection and measurement of actin in the blood and urine in patients with sepsis or sepsis-related acute kidney injury, as the early recognition of kidney injury - especially in sepsis - is essential in the aspect of therapy and survival.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* Sepsis-related acute kidney injury

Exclusion Criteria:

* malignancies needing palliative care
* end-stage renal disease
* kidney transplantation
* under 18 years of age
* unobtainable consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed septic or sepsis-related acute kidney injury patients
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Urinary actin concentrations | 3 days
  Urine samples were centrifuged (10 min, 1500 g) and supernatants were treated with electrophoresis sample buffer then heated at 100 °C for 5 minutes. Urinary actin was determined by quantitative Western blot. Native and denatured sample aliquots were stored at -70 °C until analysis.
Serum actin concentrations | 3 days
  Clotted blood samples were centrifuged (10 min, 1500 g) and supernatants were treated with electrophoresis sample buffer then heated at 100 °C for 5 minutes. Serum actin was determined by quantitative Western blot. Native and denatured sample aliquots were stored at -70 °C until analysis.

SECONDARY OUTCOMES:
U-actin/u-creatinine concentrations | 5 days
  U-actin values were determined by quantitative Western blot, while U-creatinine concentrations were measured using automated routine laboratory procedures, therefore U-actin/u-creatinine ratios could be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Dániel Ragán, MD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Péter Kustán, MD, PhD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Zoltán Horváth-Szalai, MD, PhD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Balázs Szirmay, MD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Beáta Bugyi, MD, PhD, Principal Investigator — Department of Biophysics, Medical School, University of Pécs; Andrea Ludány, MD, PhD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Attila Miseta, MD, DsC, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Bálint Nagy, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Therapy, Medical School, University of Pécs; Diána Mühl, MD, PhD, Study Director — Department of Anesthesiology and Intensive Therapy, Medical School, University of Pécs
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Medical School, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ragan D, Kustan P, Horvath-Szalai Z, Szirmay B, Bugyi B, Ludany A, Miseta A, Nagy B, Muhl D. Urinary actin, as a potential marker of sepsis-related acute kidney injury: A pilot study. PLoS One. 2021 Jul 26;16(7):e0255266. doi: 10.1371/journal.pone.0255266. eCollection 2021. PMID 34310652